CLINICAL TRIAL: NCT07298174
Title: Wide Field OCTA in Ocular Diseases: a Prospective Observational Study of the Clinical Impact of Wide Field OCTA in Ocular Disease.
Brief Title: Wide Field OCTA in Ocular Diseases
Acronym: WOOD-2025
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Alessandro Arrigo, MD, PhD, Head of Imaging Unit, Ophthalmology Department, IRCCS San Raffaele
Other Study IDs: WOOD-2025
Record Dates: First submitted 2025-12-07; First posted 2025-12-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Age - Related Macular Degeneration (AMD); Diabetic Macular Edema; Diabetic Retinopathy; Myopia; Inherited Retinal Disease; Stargardt Disease; Retinitis Pigmentosa (RP); Best Disease; Geographic Atrophy; Macular Neovascularisation; Ocular Surface Disease; Central Serous Choroidopathy; Pachychoroid Disease; Uveitis; Vitreoretinal Disease; Retinal Vein Occlusion
Keywords: wide-field octa; multimodal retinal imaging; quantitative imaging; retinal disease; macular disease; ocular surface disease
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Myopia; Stargardt Disease; Retinitis Pigmentosa; Vitelliform Macular Dystrophy; Geographic Atrophy; Central Serous Chorioretinopathy; Uveitis; Retinal Vein Occlusion; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients affected by ocular diseases: Patients affected by one of the following: AMD, diabetic retinopathy, pachychoroid spectrum, inherited retinal diseases, uveitis, ocular surface disorders

SUMMARY:
The main retinal diseases, whether or not associated with specific mutations genetic, cause progressive degeneration of vascular retinal structures and not vascular, resulting in decreased visual function. Often, such diseases affect the noblest part of the retina, called macula. Many retinal diseases can be complicated by choroidal neovascularization which causes frequent bleeding and fluid leakage that accumulates in the subretinal and intraretinal spaces. Although the investigators know many details of each disease affecting the retina, very often the correct diagnostic framework can be complicated, given the presence of morphological elements common to the different pathologies. Similarly, predicting the effect of treatment and the patient's outcome is a constant challenge for the ophthalmologists. Most of the current research has been focused on the assessment of vascular alterations localized in the macula. However, growing evidence highlight the importance of peripheral vascular changes on the outcome of retinal diseases. These changes can be detected only be wide field OCT devices.

On the other hand, ocular inflammation and hyperemia represent major assessments in anterior segment disorders, such as dry eye disease. The current grading systems of ocular inflammation, redness and hyperemia are characterized by several limitations, thus making these evaluations still mainly confined to the subjective assessment performed by the ophthalmologist. However, the new generation OCT devices may include also an anterior segment module which can reconstruct anterior segment vessels, non-invasively, using the same technology described for retinal diseases.

The main goal of the study is to evaluate the diagnostic contribution of a new generation wide field OCTA device in ocular diseases, which has recently received CE marking. In particular, the investigators will evaluate this new generation device both in retinal and anterior segments diseases, testing for common points and differences with the standard of care non-invasive diagnostic devices. Secondary outcomes include the assessment of the correlation between the patient's visual function (visual acuity) and morphological changes (standard of care imaging assessment) highlighted by the wide field OCT device, with particular attention to microstructural differences between major ocular diseases and the possible development of non-invasive biomarkers, useful for the diagnosis and follow-up of such pathologies.

DETAILED DESCRIPTION:
Hypothesis: wide field OCT may remarkably contribute on the improvement of diagnostic workup and precision medicine of ocular diseases.

Design: Post-market medical device, monocentric trial. Both cross-sectional and prospective.

The number of study groups and study duration: patients affected by ocular diseases (age-related macular degeneration, diabetic retinopathy, inherited retinal dystrophies, uveitis, myopia, pachychoroid spectrum, dry eye) and healthy controls. Duration 2-years.

the investigators will not expect remarkable biases since our evaluation will be based on the statistical analysis of quantitative imaging metrics coming from the investigational device and the comparator devices.

Both patients and controls will undergo complete ophthalmology assessment and non-invasive imaging diagnostic investigation.

In this study, the investigators will employ one standard-of-care device-Heidelberg Spectralis for retinal imaging and Keratograph 4M for anterior segment evaluation-alongside DreamOCT as the comparator device, replacing the second standard-of-care device typically used in our clinic. This is accepted and agrees with study design since, for diagnostic devices, the procedure to obtain CE approval includes safety check and comparability with other existing devices. Hence, the above described procedure represents the standard of care methodology when testing a novel device in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Both genders
* Confirmed diagnosis of one of the above diseases
* Age-related macular degeneration
* Diabetic retinopathy
* Myopia
* Pachychoroid spectrum disease
* Inherited retinal dystrophy
* Uveitis
* Dry eye
* Visual acuity of at least 1/20
* Signed informed consent for the participation to the trial.

Exclusion Criteria:

* Media opacities
* Any other eye or systemic condition that may irreversibly impair the results of the study
* Surgery in the eye in the study, including cataract extraction, in the three months prior to recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by ocular diseases and healthy controls to be considered as reference.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Retinal vessel density | Cross-sectional investigation at baseline and after 1-year follow-up
  Quantitative analysis of macular and peripheral capillary perfusion
Conjunctival vessel density | Cross-sectional investigation at baseline and after 1-year follow-up
  Conjuctival perfusion in ocular surface diseases

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available